CLINICAL TRIAL: NCT04290572
Title: Efficacy and Safety of Oral Isotretinoin 10 mg, 20 mg and 30 mg for the Treatment of Facial Recalcitrant Flat Warts at Centro Dermatológico "Dr. Ladislao de la Pascua": Randomized Double-blinded Clinical Trial of Three Arms
Brief Title: Efficacy and Safety of Oral Isotretinoin for the Treatment of Facial Recalcitrant Flat Warts
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centro Dermatológico Dr. Ladislao de la Pascua (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 176/2019
Record Dates: First submitted 2020-02-27; First posted 2020-03-02 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Flat Wart
Keywords: flat wart; isotretinoin; facial warts
MeSH Terms: interventions — Isotretinoin; Retinoids

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial of three-arms
Who Masked: Participant, Outcomes Assessor
Masking Description: All the interventions will be similar in appearance and all the participants will take the same quantity of capsules.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Isotretinoin 10 mg/day (Experimental): One capsule of isotretinoin 10 mg plus one capsule of placebo, per day during 12 weeks.
  Interventions: Drug: Isotretinoin capsules
- Isotretinoin 20 mg/day (Experimental): One capsule of isotretinoin 20 mg plus one capsule of placebo, per day during 12 weeks.
  Interventions: Drug: Isotretinoin capsules
- Isotretinoin 30 mg/day (Active Comparator): One capsule of isotretinoin 10 mg plus one capsule of isotretinoin 20 mg, per day during 12 weeks.
  Interventions: Drug: Isotretinoin capsules

INTERVENTIONS:
Drug: Isotretinoin capsules — Jelly capsules of isotretinoin
  Other Names: Oral retinoid

SUMMARY:
Randomized clinical trial to compare the efficacy of different doses of oral isotretinoin 10 mg/day, 20 mg/day and 30 mg/day during 12 weeks for the treatment of facial recalcitrant flat warts. The primary endpoint will be the proportion of participants with total remission of facial flat warts at the end of the intervention in the three arms of the clinical trial.

DETAILED DESCRIPTION:
The investigators will recruit 162 participants with facial recalcitrant flat warts and randomize to the following three arms of intervention: Arm 1: nne capsule of isotretinoin 10 mg plus one capsule of placebo, per day during 12 weeks; Arm 2: one capsule of isotretinoin 20 mg plus one capsule of placebo, per day during 12 weeks; and Arm 3: one capsule of isotretinoin 10 mg plus one capsule of isotretinoin 20 mg, per day during 12 weeks. The primary endpoints will be the proportion of participants with total remission of facial flat warts at the end of the intervention in the three arms of the clinical trial; and the incidence of side effects related to oral isotretinoin treatment among the 3 arms of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and histological diagnosis of facial flats warts
* More than 2 years with facial flat warts
* Without response to 2 or more topical interventions (tretinoin, imiquimod, cryosurgery and 5-fluorouracil) or oral interventions (cimetidine or zinc sulfate)

Exclusion Criteria:

* Have the following conditions:

  1. Hypercholesterolemia
  2. Hypertriglyceridemia
  3. Liver disease
  4. Renal disease
  5. Sjögren syndrome
  6. Pregnancy
  7. Lactation
  8. Depressive disorder
  9. Body mass index less than 18 points or higher than 25 points
  10. Contraindications for hormonal contraception or intrauterine device.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 162 (Estimated)
Dates: Start 2020-03-15 (Estimated); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete clearance | 12 weeks
  Proportion of participants with total remission of facial flat warts at the end of the intervention in the three arms of the clinical trial.
Incidence of serious adverse events | 12 weeks
  Proportion of participants that developed a serious side effect in the three arms during the clinical trial.

SECONDARY OUTCOMES:
Quality of life index | 12 weeks
  Difference in the Dermatology Life Quality Index score at the end of the study, comparing with the basal score. The minimum score is 0 points and the maximum 30 points. A score higher than 10 points means that the patient's life is severely affected by melasma.
Adherence to intervention | 12 weeks
  Percentage of taken-doses of oral isotretinoin during the 12 weeks of the study.

CONTACTS AND LOCATIONS:
Overall Officials: María Guadalupe Olguín-García, M.D.,MSc., Principal Investigator — Centro Dermatológico Dr. Ladislao de la Pascua
Locations (1):
- Centro Dermatológico "Dr. Ladislao de la Pascua", Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No